CLINICAL TRIAL: NCT04883827
Title: Monitoring Disease Burden and Biology Using Tumor Cell Free DNA in Metastatic Kidney Cancer
Brief Title: Disease Burden and Biology Using Tumor Cell Free DNA in Metastatic Kidney Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott Haake, MD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC URO 2144
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RCC with clear cell component
  Interventions: Other: Blood collection; Other: Urine collection
- Healthy Volunteer (no longer recruiting)
  Interventions: Other: Blood collection; Other: Urine collection

INTERVENTIONS:
Other: Blood collection — 20-40 mL of blood to extract cell free DNA
Other: Urine collection — up to 15 mL of urine to extract cell free DNA

SUMMARY:
This study will assess whether DNA released by kidney cancer into the blood stream and urine of patients can be used to monitor tumor burden and tumor response to treatment in patients receiving immunotherapy

DETAILED DESCRIPTION:
Primary Objective:

- Evaluate tumor cell free (cf)DNA as a dynamic marker of response to immuno-oncology (IO) therapy

Exploratory Objective:

- Collect data on somatic mutations in cfDNA to gain insight into the biology of IO-responders and -non-responders

ELIGIBILITY:
Inclusion Criteria:

* Renal Cell Carcinoma with clear cell component
* Stage IV
* Receiving IO-containing regimen
* Measurable disease per RECIST 1.1

Exclusion Criteria:

* Active cancer (exclusion criteria only for healthy patient cohort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (18 year or older) with Renal Cell Carcinoma with clear cell component and receiving an IO-containing regimen or healthy volunteers (18 years or older)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluate tumor cfDNA as a dynamic marker of response to IO therapy | Up to about 2 years
  Measure of changes in the amount of tumor DNA correlated with result of routine tumor imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Scott Haake, MD, Principal Investigator — Vanderbilt Medical Center
Locations (3):
- United States (3):
  - Tennessee Valley Health Care System, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT04883827/ICF_000.pdf